CLINICAL TRIAL: NCT03939845
Title: A Prospective, Randomized, Multicenter Study of Comparison of Transarterial Chemoembolization (TACE) Combination With and Without External- Beam Radiotherapy (EBRT) for Hepatocellular Carcinoma With Portal Vein Tumor Thrombi
Brief Title: A Prospective, Randomized, Multicenter Study of Comparison of TACE Combination With and Without EBRT for Hepatocellular Carcinoma With Portal Vein Tumor Thrombi
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PVT/RT
Record Dates: First submitted 2019-04-23; First posted 2019-05-07 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-04

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TACE (Active Comparator)
  Interventions: Procedure: TACE
- TACE+RT (Experimental)
  Interventions: Radiation: RT; Procedure: TACE

INTERVENTIONS:
Radiation: RT — external- beam radiotherapy (EBRT)
  Arms: TACE+RT
Procedure: TACE — transarterial chemoembolization (TACE)

SUMMARY:
The 1-year and 2-year overall survival rate (OS), local control rate (FFLP), disease-free progression time (PFS), and side effects were compared in patients with hepatocellular carcinoma limited to intrahepatic unresectable hepatocellular carcinoma with portal venous thrombosis combined with or without external radiotherapy, providing a basis for the development of relevant guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed by pathology or met the clinical diagnostic criteria of hepatocellular carcinoma.
2. after the joint consultation between the interventional department and the radiotherapy department, the patients who were considered to be interventional were considered. Meeting the following criteria: the tumor was confined to the liver (meeting the liver tolerance dose), and was diagnosed as type II or type III portal vein tumor thrombi according to chang's classification criteria, without extrahepatic metastasis. Number of tumors in liver parenchyma: less than or equal to 3. The main portal vein is not completely blocked or the compensatory collateral vessels of the portal vein are abundant although it is completely blocked.
3. patients who meet all the following criteria: Child-Pugh score ≤7, PLT>30×109/L, WBC>3×10^9/L/ANC>1.5×10^9/L,Hb>90g/L, Cr<2.0mg/dL.
4. ECOG score 0-2 points.
5. estimated survival time > 3 months.
6. age > 18.
7. sign the informed consent.

Exclusion Criteria:

1. patients with the following condition: the number of intrahepatic tumors >3 or total tumor diameter>15cm.
2. patients with signs of extrahepatic metastasis, including but not limited to inferior vena cava carcinoma thrombus, bone metastasis, brain metastasis or regional lymph node metastasis.
3. patients with West Haven standard grade III/IV hepatic encephalopathy or ascites.
4. patients with a history of malignancy other than primary HCC, except for cutaneous squamous cell carcinoma or basal cell carcinoma.
5. patients with a history of upper abdominal radiotherapy.
6. in the radiotherapy plan, patients who failed to follow the radiation dose limit of important organs, including those whose normal liver tissue was less than 700 ml in the radiotherapy plan.
7. screening patients who have received other study drugs within 4 weeks prior to the start of the visit.
8. screening: patients who had received treatment for other local or systemic hepatocellular carcinoma within 4 weeks before the visit.
9. patients with significant concurrent diseases.
10. lactating or pregnant female patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-04-23 (Estimated); Study Completion 2022-04-23 (Estimated)

PRIMARY OUTCOMES:
OS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hosptial, Shanghai, Shanghai Municipality, China